CLINICAL TRIAL: NCT00001385
Title: Positron Emission Tomography in Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940151; 94-C-0151
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Breast Neoplasms
Keywords: Cancer Diagnosis; Cancer Metabolism; FDG; FDG Breast Imaging; PET; Positron Emission Mammography; Radiopharmaceutical; Scintimammography
MeSH Terms: conditions — Breast Neoplasms

SUMMARY:
This is a prospective study evaluating the role of Positron Emission Tomography (PET scan) in breast cancer. The radiopharmaceutical [18F] 2-deoxyglucose will be used as both an imaging modality and to evaluate tumor metabolism in patients with breast cancer. Patients with stage II, stage IIIA or IIIB, or stage IV breast cancer and evaluable disease in the breast and/or at metastatic sites will be studied. Patients will be injected intravenously with [18F]2-deoxyglucose and a PET scan conducted over 90 minutes. Examination of the role of PET scan in assessing the response of breast cancer to chemotherapy, especially in stage II and stage III patients, will be done. Up to three PET scans within one year may be performed. Findings by PET scan will be correlated both with those of concurrent imaging techniques (x-ray, CT scan, MRI, bone scan or mammogram), and with histologic, biochemical, and flow cytometric information on the tumor, and with findings in subsequent surgical specimens. Changes in tumor glucose metabolism with treatment will be assessed by PET imaging studies and by biochemical methods when possible.

DETAILED DESCRIPTION:
This is a prospective study evaluating the role of Positron Emission Tomography (PET scan) in breast cancer. The radiopharmaceutical [18F] 2-deoxyglucose will be used as both an imaging modality and to evaluate tumor metabolism in patients with breast cancer. Patients with stage II, stage IIIA or IIIB, or stage IV breast cancer and evaluable disease in the breast and/or at metastatic sites will be studied. Patients will be injected intravenously with [18F]2-deoxyglucose and a PET scan conducted over 90 minutes. Examination of the role of PET scan in assessing the response of breast cancer to chemotherapy, especially in stage II and stage III patients, will be done. Up to three PET scans within one year may be performed. Findings by PET scan will be correlated both with those of concurrent imaging techniques (x-ray, CT scan, MRI, bone scan or mammogram), and with histologic, biochemical, and flow cytometric information on the tumor, and with findings in subsequent surgical specimens. Changes in tumor glucose metabolism with treatment will be assessed by PET imaging studies and by biochemical methods when possible.

ELIGIBILITY:
Histologically proven invasive carcinoma of the breast.

Patients with stage II, stage IIIA or IIIB, or stage IV breast cancer who have not received local therapy to the breast or axillary lymph nodes.

Evaluable tumor, either gross or microscopic, at locoregional and/or distant sites.

No current pregnancy.

No second invasive malignancy in addition to breast cancer.

No significant concurrent medical disorders (cardiac, renal, hepatic).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 1994-05; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wahl RL, Cody RL, Hutchins GD, Mudgett EE. Primary and metastatic breast carcinoma: initial clinical evaluation with PET with the radiolabeled glucose analogue 2-[F-18]-fluoro-2-deoxy-D-glucose. Radiology. 1991 Jun;179(3):765-70. doi: 10.1148/radiology.179.3.2027989.
- [Background] Di Chiro G, Brooks RA. PET-FDG of untreated and treated cerebral gliomas. J Nucl Med. 1988 Mar;29(3):421-3. No abstract available. PMID 3258029